CLINICAL TRIAL: NCT02390492
Title: A Phase I Study to Investigate the Absorption, Metabolism, and Excretion of [14C]-Ipatasertib (GDC-0068) Following a Single Oral Dose and to Investigate the Absolute Bioavailability Following Single Oral and Intravenous Doses in a Single Cohort of Healthy Male Subjects
Brief Title: A Phase I Bioavailability and Pharmacokinetic Study of [14C]-Ipatasertib Single Oral and Intravenous Doses in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: GP29067
Record Dates: First submitted 2015-03-11; First posted 2015-03-17 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer

ARMS (1):
- Ipatasertib/[14C]-ipatasertib (Experimental)
  Interventions: Drug: Period 1 treatment; Drug: Period 2 treatment

INTERVENTIONS:
Drug: Period 1 treatment — 200 mg oral ipatasertib followed 1 hour later by 80-mcg/800-nCi intravenous [14C]-ipatasertib on Day 1 of study
Drug: Period 2 treatment — 200-mg/100-mcCi oral [14C]-ipatasertib on Day 15 of study

SUMMARY:
This 2-period, open-label, nonrandomized study will be conducted to determine the absolute bioavailability as well as the absorption, metabolism, and excretion of ipatasertib and its metabolite(s). Healthy male participants will receive a single 200-mg oral dose of ipatasertib followed 1 hour later by an 80-mcg/800-nCi intravenous dose of [14C]-ipatasertib. After a 4-day observation period and 10-day washout, participants will receive a single 200-mg/100-mcCi oral dose of [14C]-ipatasertib with subsequent data collection for an additional 7 to 14 days until discharge criteria are met.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers 18 to 55 years of age, inclusive
* Body mass index (BMI) 18 to 32 kg/m2, inclusive

Exclusion Criteria:

* Females
* Clinically significant findings from medical history or screening evaluations
* Recent participation in any other investigational drug study or biologic agent study, or receipt of a previous radiolabeled investigational drug within 6 months prior to check-in
* Significant radiation exposure within 12 months prior to check-in

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2015-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of [14C]-ipatasertib/ipatasertib (oral): apparent terminal elimination half-life | Period 2: Approximately 2 weeks
Pharmacokinetics of ipatasertib (oral): apparent total clearance (CL/F) | Period 2: Approximately 2 weeks
Pharmacokinetics of ipatasertib (oral): apparent volume of distribution (Vz/F) | Period 2: Approximately 2 weeks
Elimination and pharmacokinetics: Total radioactivity concentration in whole blood, plasma, urine, and feces | Period 2: Approximately 2 weeks
Bioavailability: Absolute bioavailability of ipatasertib (area under the concentration-time curve) | Period 1: Approximately 4 days
Mass balance | Period 2: Approximately 2 weeks
Pharmacokinetics of [14C]-ipatasertib/ipatasertib (oral): maximum observed concentration (Cmax) | Period 2: Approximately 2 weeks
Pharmacokinetics of [14C]-ipatasertib/ipatasertib (oral): time to maximum observed concentration (Tmax) | Period 2: Approximately 2 weeks
Pharmacokinetics of [14C]-ipatasertib/ipatasertib (oral): area under the concentration-time curve from Hour 0 to the last measurable concentration (AUC0-t) | Period 2: Approximately 2 weeks
Pharmacokinetics of [14C]-ipatasertib/ipatasertib (oral): area under the concentration-time curve extrapolated to infinity (AUC0-inf) | Period 2: Approximately 2 weeks
Pharmacokinetics of [14C]-ipatasertib/ipatasertib (oral): apparent terminal elimination rate constant | Period 2: Approximately 2 weeks

SECONDARY OUTCOMES:
Pharmacokinetics of ipatasertib (oral and IV): terminal elimination rate constant adjusted for oral bioavailability as applicable | Period 1: Approximately 4 days
Pharmacokinetics of ipatasertib (oral and IV): terminal elimination half-life adjusted for oral bioavailability as applicable | Period 1: Approximately 4 days
Pharmacokinetics of ipatasertib (oral and IV): total clearance adjusted for oral bioavailability as applicable | Period 1: Approximately 4 days
Pharmacokinetics of ipatasertib (oral and IV): volume of distribution adjusted for oral bioavailability as applicable | Period 1: Approximately 4 days
Safety: Incidence of adverse events | Approximately 4 weeks
Elimination and pharmacokinetics: Metabolite concentration(s) in plasma, urine, and feces | Period 2: Approximately 2 weeks
Pharmacokinetics of ipatasertib (oral and IV): Cmax | Period 1: Approximately 4 days
Pharmacokinetics of ipatasertib (oral and IV): Tmax | Period 1: Approximately 4 days
Pharmacokinetics of ipatasertib (oral and IV): AUC0-t | Period 1: Approximately 4 days
Pharmacokinetics of ipatasertib (oral and IV): AUC0-inf | Period 1: Approximately 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Madison, Wisconsin, United States